CLINICAL TRIAL: NCT05913973
Title: Phase 1 Dose Escalation Study of The Plasmodium Vivax Transmission-Blocking Vaccine Pvs230D1-EPA/Matrix-M to Assess Safety, Immunogenicity, and Transmission-Blocking Activity in Healthy Malaria-Naive Adults
Brief Title: Study of the Plasmodium Vivax Transmission-blocking Vaccine Pvs230D1-EPA/Matrix-M to Assess Safety, Immunogenicity, and Transmission-blocking Activity in Healthy Malaria-naive Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 10001501; 001501-I
Record Dates: First submitted 2023-06-19; First posted 2023-06-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11-26

CONDITIONS: Malaria
Keywords: TBV; Open Label; Antibody; Reactogencity; Mosquito
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): 5 (micro)g Pvs230D1-EPA/50 (micro)g MM
  Interventions: Drug: Pvs230D1-EPA/Matrix-M
- Group 2 (Experimental): 25 (micro)g Pvs230D1-EPA/50 (micro)g MM
  Interventions: Drug: Pvs230D1-EPA/Matrix-M
- Group 3 (Experimental): 50 (micro)g Pvs230D1-EPA/50 (micro)g MM
  Interventions: Drug: Pvs230D1-EPA/Matrix-M

INTERVENTIONS:
Drug: Pvs230D1-EPA/Matrix-M — Pvs230 domain 1 (Pvs230D1) is a recombinant protein consisting of subdomain 1 of native Pvs230 (Val-226 to Gly-427, Figure 2) produced in Pichia pastoris. The synthetic gene sequence was optimized for P. pastoris expression and cloned into the expression vector pPICZ(alpha)A, which also encodes a pre-prosecretory alpha-factor sequence.

SUMMARY:
Background:

Malaria is a disease carried by mosquitoes in tropical countries around the world. It can cause symptoms like fever, body aches, and weakness. More than half a million people worldwide died of malaria in 2021, mostly children. Researchers want to find ways to prevent the spread of this disease.

Objective:

To test the effects of a new malaria vaccine. (Volunteers will not be exposed to malaria.)

Eligibility:

Healthy adults aged 18 to 50 years.

Design:

Volunteers will be screened. They will have a physical exam with blood and urine tests. They will take a short quiz to make sure they understand the study.

Volunteers will have 3 visits to receive the vaccine. These visits will be about 1 month apart. The vaccine will be injected into the muscle of the upper arm.

Volunteers will have 12 additional clinic visits. These will start after the first vaccine visit and continue for 8 months. The visits may include a physical exam and blood tests. There will also be 7 follow-up phone calls. These will occur the day after each vaccine visit and then continue for another 12 months. Participants will be asked how they are doing and whether they have had any changes in their health.

...

DETAILED DESCRIPTION:
Study Description:

Single-center, open-label, first-in-human, dose-escalating phase 1 study to characterize the safety, immunogenicity, and transmission-blocking activity in healthy malaria-naive adults of the Plasmodium vivax (P. vivax) transmission-blocking vaccine (TBV), Pvs230D1-EPA combined with adjuvant Matrix-M (MM). Three doses of vaccine will be administered at 1-month intervals (study days 0, 28, and 56). Subjects will be divided into low, intermediate, and high dose groups based on the amount of the antigen component in each vaccine dose:

* Group 1 (n = 10): 5 (micro)g Pvs230D1-EPA/50 (micro)g MM
* Group 2 (n = 10): 25 (micro)g Pvs230D1-EPA/50 (micro)g MM
* Group 3 (n = 10): 50 (micro)g Pvs230D1-EPA/50 (micro)g MM

Objectives:

Primary Objective

-To assess the safety and reactogenicity of Pvs230D1-EPA/MM in healthy malaria-naive adults

Exploratory Objectives

* To determine the antibody response to Pvs230D1-EPA/MM
* To determine the functional response to Pvs230D1-EPA/MM by mosquito feeding assays
* To assess cellular and transcriptomic responses to Pvs230D1-EPA/MM
* To identify and characterize human monoclonal antibodies (mAbs) with activity against Pvs230D1M

Endpoints:

Primary Endpoint

-Incidence and severity of local and systemic adverse events (AEs) or serious adverse events (SAEs)

Exploratory Endpoints

* Anti-Pvs230D1M antibody levels as measured by enzyme-linked immunosorbent assay (ELISA)
* Transmission-reducing activity (TRA) and/or transmission-blocking activity (TBA) of Pvs230D1-EPA/MM using direct membrane feeding assays (DMFA)
* Cellular immune responses and whole genome transcriptional profiles
* Isolation of reactive antibodies from sorted B cells

ELIGIBILITY:
* INCLUSION CRITERIA:

All of the following criteria must be fulfilled for a subject to participate in this trial:

1. Age >=18 and <=50 years.
2. In good general health and without clinically significant medical history.
3. Able to sign a written informed consent prior to undertaking any study-related procedure.
4. Vaccine comprehension exam completed, passed (a score of (Bullet)80% or per investigator s discretion), and reviewed prior to enrollment.
5. Suitable accommodation and reliable access to the NIHCC for the duration of the study, in the opinion of the investigator.
6. Individuals of childbearing potential must agree to use an acceptable method of contraception from 1 month prior to enrollment to 1 month after the final vaccination (i.e., from study day -28 until study day 84).
7. Individuals capable of fathering children must agree to use an acceptable method of contraception from 1 month prior to enrollment to 1 month after the final vaccination (i.e., from study day -28 until study day 84).
8. Willing to allow long-term storage of study samples for future research.
9. Willing to refrain from donating blood throughout the study until 6 months after the last vaccination.

EXCLUSION CRITERIA:

A subject will be excluded from participating in this trial if any 1 of the following criteria is fulfilled:

1. Planned travel to a malaria-endemic area until 6-months beyond the final vaccination (see https://www.cdc.gov/malaria/travelers/country_table/a.html). Exceptions may be made, at the investigator s discretion, if the travel is limited to areas without appreciable levels of P. vivax transmission.
2. Any prior confirmed P. vivax malaria diagnosis or clinical history consistent with P. vivax malaria diagnosis within the previous 10 years, at the investigator's discretion.
3. Any subject without good peripheral venous access, at the investigator's discretion.
4. For individuals of childbearing potential:

   1. Currently breastfeeding.
   2. Currently pregnant as determined by history or a positive human choriogonadotropin (beta-hCG) test.
5. Clinical trial staff with direct involvement in the conduct of the trial are excluded from participation.
6. HIV, hepatitis B, and/or hepatitis C as determined by HIV antigen/antibody, Hepatitis B surface antigen, and anti-Hepatitis C antibody laboratory tests.
7. Screening blood test or urinalysis laboratory parameters outside of local lab normal range. Subjects may be included at the investigator s discretion for "not clinically significant" values outside of normal range.
8. History of anaphylaxis, severe allergy, or other concerning adverse reaction, in the opinion of the investigator, to a previous vaccine.
9. Any of the following within the specified periods:

   1. Investigational P. vivax malaria vaccine within the last 2 years.
   2. Chronic systemic immunosuppressive medications (>14 days) within 6 months of study day 0 (e.g., cytotoxic medications, adrenocorticotrophic hormone, or oral/parental corticosteroids equivalent to >0.5 mg/kg/day of prednisone). Corticosteroid nasal spray for allergic rhinitis and topical corticosteroids for mild, uncomplicated dermatitis are allowed at the discretion of the investigator.
   3. Investigational or non-FDA approved/authorized product or vaccine within 28 days prior to study day 0.
   4. Asplenia or functional asplenia.
   5. Blood transfusion or IVIG within 6 months of study day 0.
10. Any other finding that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a subject s ability to give informed consent, or increase the risk of having an adverse outcome from participating in the study.

Subjects who are excluded from participation for any of the reasons above may be considered for

enrollment on a postponed schedule if the investigator considers this appropriate.

Subjects will be selected in an equitable manner from the available pool of potentially eligible individuals, without regard to factors such as sex, gender, race, ethnicity, socioeconomic status, etc., except for age.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety and reactogenicity of Pvs230D1-EPA/MM in healthy malaria-naive adults | Receipt of first vaccine through subject study completion
  Incidence and severity of local and systemic adverse events (AEs) or serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Joel A Goldberg, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This study will be conducted in accordance with the following publication and data sharing policies and regulations:@@@@@@NIH Public Access Policy, which ensures that the public has access to the published results of NIH funded research. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive PubMed Central upon acceptance for publication.@@@@@@This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals. @@@@@@

REFERENCES:
- [Derived] Cao Y, da Silva Araujo M, Lorang CG, Dos Santos NAC, Tripathi A, Vinetz J, Kumar N. Distinct immunogenicity outcomes of DNA vaccines encoding malaria transmission-blocking vaccine target antigens Pfs230D1M and Pvs230D1. Vaccine. 2025 Feb 15;47:126696. doi: 10.1016/j.vaccine.2024.126696. Epub 2025 Jan 8. PMID 39787798
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001501-I.html